CLINICAL TRIAL: NCT00232349
Title: An Open-Label Trial of Adjunctive Galantamine Maintenance Therapy to Treat Functional Impairments in Chronic Outpatients With Schizophrenia
Brief Title: Efficacy of Galantamine to Treat Schizophrenia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to no apparent benefit.
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Responsible Party: Andre Tapp, M.D., VA Puget Sound Health Care System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA1 28; GAL-EMR-4009
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2008-07-31 (Estimated); Status verified 2008-07

CONDITIONS: Schizophrenia; Psychotic Disorder
Keywords: schizophrenia; galantamine; cholinesterase inhibitors; quality of life; cognition
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Galantamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention group (Experimental): All subjects enrolled in study are in the intervention group.
  Interventions: Drug: galantamine

INTERVENTIONS:
Drug: galantamine — open label galantamine, dosed at 4-12 mg/b.i.d., with a target dose of 12 mg/b.i.d.
  Other Names: Razadyne; Reminyl

SUMMARY:
The purpose of this study was to determine if treatment with adjunctive galantamine is effective in the reduction of functional impairments in patients with schizophrenia and schizoaffective disorder. It was hypothesized that adjunctive galantamine would yield clinically significant improvements from baseline to end of study on a measure of quality of life and a measure of independent living skills.

DETAILED DESCRIPTION:
A majority of patients with schizophrenia or schizoaffective disorder experience impairments in social relations and employment. Many patients experience impairments in their ability to live independently, requiring assistance in such activities as money management, shopping, food preparation and hygiene. These impairments in functioning have been shown to be related to cognitive deficits associated with the disease.

Galantamine is a medication that has been approved by the FDA for the treatment of mild to moderate Alzheimer's disease. Both animal and human models have shown that galantamine can enhance learning and memory. Case reports and preliminary research have suggested that galantamine is an effective adjunctive treatment for schizophrenia, improving both cognition and negative symptoms. Improvements in functioning require that gains in cognition be maintained long enough to allow for the acquisition and application of new skills and behaviors.

Thus, this nine month, open label study assessed the efficacy of galantamine, dosed at 4-12 mg/twice a day, for the treatment of functional impairments in individuals, ages 18-60, with schizophrenia and schizoaffective disorder. The primary outcome measures were changes from baseline to end of study in scores on the Independent Living Scale (ILS) and the Quality of Life Scale (QLS). Secondary outcome measures included assessments of symptoms, cognition, side effects, and movement disorders.

Twenty-one subjects signed informed consent and fourteen subjects were initiated on medication. Six subjects completed the study. As per a priori plan, those subjects (n = 8) who were treated with study medication for at least four months were included in the analyses of treatment outcomes. Our findings regarding the efficacy of galantamine for functional outcomes, including activities of daily living and quality of life, did not support our hypothesis that long-term treatment with galantamine would yield improvements in these domains in patients with schizophrenia spectrum disorders. In fact, in the current study, we did not observe any anticipated improvements in cognition. In addition, we did not observe any anticipated improvements in symptoms, specifically negative symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* Able to provide informed, written consent
* Treatment for schizophrenia or schizoaffective disorder for 5 or more years
* Diagnosis of schizophrenia or schizoaffective disorder
* Psychiatrically stable as evidenced by no hospitalizations and no changes in psychiatric medications (with the exception of dosage adjustments and the prescription of adjunctive treatments for sleep disturbance or anxiety) within the prior 3 months, and as confirmed by clinical interview during the screening phase
* Total score > 60 baseline on The Positive and Negative Syndrome Scale (PANSS)
* Score > 3 on at least one of the five subscales of the SANS
* Non-Kraepelinian schizophrenia, as defined by the ability to independently provide for at least one domain of basic needs
* Females must be of non-child bearing potential or on appropriate contraceptive and not breast-feeding
* Females must have a negative serum beta HCG at screening
* Clinical laboratory values within normal limits, as defined in study protocol, or abnormalities considered not clinically significant by the investigator

Exclusion Criteria:

* Kraepelinian schizophrenia, as defined by dependency on others for the provision of all basic needs (including shopping, food preparation, household chores, and transportation);
* DSM-IV criteria for substance dependence (excluding nicotine and caffeine), as determined by SCID and chart review, during the 90 days prior to screening;
* Patients judged by the investigator as being at significant risk of suicide, violent behavior, or homicide;
* Concurrent participation or participation within the prior 30 days in any study involving investigational medications;
* Females who are pregnant or lactating;
* Neurodegenerative disorders such as Alzheimer's disease and other dementias, Parkinson's disease, Pick's disease, and Huntington's chorea;
* A history of significant cerebrovascular event yielding a physical or neurological deficit likely to confound the assessment of the subject's functioning;
* A history of significant head trauma, defined as head trauma resulting in neurological or cognitive sequelae;
* A known personal history of seizure disorder;
* A known sensitivity to cholinesterase inhibitors, choline agonists, or similar agents;
* Patients who are known to be HIV positive;
* Evidence of clinically significant, active gastrointestinal, hepatic, pulmonary, endocrine, renal, or cardiovascular system disease;
* Active or clinically significant conditions affecting absorption, distribution or metabolism of the study medication (e.g. inflammatory bowel disease or gastric or duodenal ulcers);
* Clinically significant urinary outflow obstruction;
* Patients with untreated thyroid disease;
* Patients with Type I or Type II diabetes controlled by medication or diet who do not have a HbA1c of < 8.5%;
* Patients with known significant cardiac history such as myocardial infarction or abnormal cardiac catheterization within the last 12 months.
* Unstable angina: angina or coronary artery disease requiring a change in medications within the 3 months prior to screening;
* Decompensated congestive heart failure;
* Severe mitral or aortic valvular disease;
* Atrial fibrillation;
* Greater than first degree atrioventricular block;
* QTc prolongation at screening;
* Bradycardia <50 beats/min;
* Current treatment with clozapine, olanzapine, chlorpromazine, or thioridazine;
* Use of potent cytochrome P450 inhibitors or inducers within 14 days before the Baseline Visit or during treatment, as listed in Appendix B of protocol;
* Current use of potent anticholinergic medication, as listed in Appendix B;
* Current use of any disallowed concomitant medication, as listed in Appendix B; and
* Any clinical finding that in the opinion of the investigator could potentially be negatively affected by study participation or that could potentially affect study participation is criterion for exclusion from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2005-02; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
score on a measure of quality of life | after 9 months treatment
score on a measure of independent living skills | after 9 months treatment

SECONDARY OUTCOMES:
score on a measure of psychopathology | after 9 months treatment
score on a measure of negative symptoms | after 9 months treatment
score on a neurocognitive battery | after 9 months treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andre Tapp, M.D., Principal Investigator — VA Puget Sound Health Care System, Tacoma and Seattle, WA and University of Washington, Department of Psychiatry and Behavioral Sciences, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System, American Lake Division, Tacoma, Washington, United States

REFERENCES:
- [Background] Allen TB, McEvoy JP. Galantamine for treatment-resistant schizophrenia. Am J Psychiatry. 2002 Jul;159(7):1244-5. doi: 10.1176/appi.ajp.159.7.1244. No abstract available. PMID 12091212